CLINICAL TRIAL: NCT03790449
Title: Evaluation of a Mobile Preconception Lifestyle Programme in Couples Undergoing in Vitro Fertilisation: a Multicentre Randomized Controlled Trial (PreLiFe-RCT)
Brief Title: Evaluation of a Mobile Preconception Lifestyle Programme in Couples Undergoing In Vitro Fertilisation
Acronym: PreLiFe-RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the worldwide Covid-19 pandemic, all Belgian fertility clinics stopped offering IVF as of March 13th 2020. We had to stop recruitment and follow-up of study subjects. We therefore adjusted our primary outcome to time to ongoing pregnancy.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: s61596
Record Dates: First submitted 2018-11-12; First posted 2018-12-31 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Infertility
Keywords: Infertility; Lifestyle; mobile health; Diet; Physical Activity; Mindfulness
MeSH Terms: conditions — Infertility; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (1:1)
Masking Description: Statistician is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PreLiFe-programme (Experimental): A Mobile Preconception Lifestyle programme
  Interventions: Behavioral: PreLiFe-programme; Behavioral: Attention Control Programme
- Attention Control (Other): Attention Control Programme
  Interventions: Behavioral: Attention Control Programme

INTERVENTIONS:
Behavioral: PreLiFe-programme — The intervention group will receive a mobile preconception lifestyle programme (the PreLiFe-programme) in addition to standard care for 12 months or until an ongoing pregnancy is confirmed by ultrasound. The PreLiFe-programme includes a mobile application (PreLiFe-app) with the same treatment information as the attention control group in combination with a lifestyle programme. This new lifestyle programme includes tailored advice and skills training on diet and physical activity and mindfulness exercises. Additionally couples will be offered interaction with a health care provider through text messages and telephone interaction following the concept of blended care.
  Arms: PreLiFe-programme
Behavioral: Attention Control Programme — The standard care serving as control for this intervention is fertility treatment i.e. IVF with or without ICSI according to local protocols for infertility patients. This implies no guidance on lifestyle. However, to have attention control the control group will receive an attention control programme. The attention control programme includes a mobile application (app) with treatment information including medication instructions, reminders of injection of human Chorionic Gonadotropin (hCG) and time of fertility treatment appointments for 12 months or until an ongoing pregnancy is confirmed by ultrasound.

SUMMARY:
The aim of the PreLiFe RCT is to assess the effects of a new mobile preconception lifestyle programme (PreLiFE-programme) for couples undergoing IVF. Couples about to start IVF will be randomized between an attention control programme or the PreLiFe-programme for 12 months or until an ongoing pregnancy is confirmed by ultrasound.This study will examine whether the PreLiFe-programme results in a higher cumulative ongoing pregnancy rate within 12 months as compared to an attention control programme. Secondary outcomes include changes in diet, physical activity, personal wellbeing, body mass index, waist circumference, quality of life and other reproductive outcomes including clinical pregnancy and time to pregnancy. Additionally, the partners' support and the feasibility of the PreLiFe-programme will be evaluated.

DETAILED DESCRIPTION:
Introduction: Infertility and in vitro fertilization (IVF; with or without intracytoplasmic sperm injection, ICSI) result in considerate emotional and financial burden. Increasing evidence suggests that lifestyle factors, including diet, physical activity and personal wellbeing, are associated with IVF-success rates. So far, IVF is not routinely combined with a lifestyle programme. The PreLiFe randomized controlled trial (RCT) will assess the effects of a new mobile preconception lifestyle programme (PreLiFe-programme) in couples undergoing IVF.

Methods and analysis: A multicentre RCT will include heterosexual couples about to start IVF (with or without ICSI) in Belgian fertility clinics. IVF-Couples will be randomized between an attention control programme or the PreLiFe-programme for 12 months or until an ongoing pregnancy is confirmed by ultrasound. The attention control programme includes a mobile application with treatment information (i.e. appointments and medication instructions) in addition to standard care. The PreLiFe-programme includes a mobile application with the same treatment information in combination with a lifestyle programme. This new lifestyle programme includes tailored advice on diet and physical activity and mindfulness exercises in combination with text messages and telephone interaction with a lifestyle coach. The primary outcome of this RCT is the cumulative ongoing pregnancy rate within 12 months after randomisation. Secondary outcomes include changes in diet, physical activity, personal wellbeing, body mass index, waist circumference and quality of life measured with self-reported questionnaires and physical assessments and changes in other reproductive outcomes including clinical pregnancy and time to pregnancy. Additionally, the partners' support and the feasibility (use and acceptability) of the PreLiFe-programme will be evaluated using self-reported questionnaires and app-based tracking. Analysis will be according to intention to treat.

Ethics and dissemination: This study has been approved by the Medical Ethical Committee of the Leuven University Hospital (Belgium) and of the other recruiting clinics. The findings of this RCT will be disseminated through presentations at international scientific meetings and peer-reviewed publications.

Due to the worldwide Covid-19 pandemic, we had to stop recruiting new patients and stop studying patients who were in the midst of their 12 months study period. This was inevitable as all Belgian fertility clinics stopped offering IVF as of March 13th 2020 for a (not predefined) period. Patients who had been randomized, but were still ongoing in the trial at that time needed to be censored. Based on statistical advise, we changed therefore our primary outcome analysis from cumulative ongoing pregnancy rate within 12 months after randomisation to time to ongoing pregnancy in order to be able to use the data of the many study patients who were in the midst of their 12 months study period.

ELIGIBILITY:
Inclusion Criteria:

* Infertile heterosexual couples about to start a first IVF-cycle (with or without ICSI) with infertility defined as the failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse
* Women of couples aged ≤ 38 years
* Both partners possess a smartphone
* Both partners understand and speak Dutch
* Written informed consent after been informed on all aspects of the study

Exclusion Criteria:

* Couples with previous IVF/ICSI treatment cycles
* Couples where one of the partners has special dietary requirements including but not limited to patients that underwent bariatric surgery, patients with coeliac disease or renal disease
* Couples where one of the partners has specific movement's constraints including but not limited to patients with cerebral palsy or hemiparesis
* Couples starting IVF/ICSI with preimplantation genetic diagnosis (PGD)
* Couples using donor gametes or donor embryos

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Cumulative ongoing pregnancy rate (COPR) within 12 months after randomisation | 12 months
  Ongoing pregnancy is defined as a viable intrauterine pregnancy of at least 12 weeks duration confirmed on ultrasound scan. All pregnancies (Spontaneous and IVF pregnancies) conceived within these 12 months are followed up until the 12 weeks ultrasound scan. IVF-discontinuation is described as couples undergoing IVF who do not return for a further IVF cycle in our fertility centres after the failure of a previous cycle. Ongoing pregnancy within 12 months after randomisation is counted as a positive event, whereas IVF discontinuation and absence of pregnancy are counted as a negative event. Differences in COPR will be evaluated between the intervention and attention control group.

SECONDARY OUTCOMES:
Changes in diet assessed with a Food Frequency Questionnaire (FFQ) | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  A validated food frequency questionnaire (FFQ) is used to evaluate changes in dietary pattern and diet quality over time and to evaluate differences in the dietary pattern and diet quality between the intervention and attention control group. The FFQ consists of a finite list of foods and beverages with response categories to indicate usual frequency and portion size of consumption over the last month. Diet quality is calculated from the FFQ by assessing quality, balance and variety of foods and beverages consumed (score 0-100 with the higher the better diet quality). Diet quality is an index to reflect compliance with the Belgian Food Based Dietary Guidelines.
Changes in physical activity assessed with the International Physical Activity Questionnaire (IPAQ) | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) is used to evaluate changes in physical activity over time and to evaluate differences in physical activity between the intervention and attention control group. The IPAQ-SF assesses the duration (in minutes) and frequency (in days) of walking, moderate-intensity activities, vigorous-intensity activities and sedentary activity (sitting) based on metabolic equivalent (MET) values. Self-reported physical activity is classified as low, moderate or high physically active based on the global recommendations on physical activity for health of the World Health Organisation. The IPAQ-SF is a reliable and validated instrument for monitoring physical activity in population health surveillance systems.
Changes in symptoms of emotional distress, anxiety and depression (personal wellbeing) assessed with the Depression, anxiety and stress scale (DASS-21) | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  The Depression, anxiety and stress scale (DASS-21) is used to evaluate changes in personal wellbeing over time and to evaluate differences in personal wellbeing between the intervention and attention control group. Self-reported symptoms of stress, anxiety and depression (together emotional distress) are measured with this validated scale (score 0-126 with the lower, the higher personal wellbeing).
Changes in fertility related quality of life assessed with the Fertility Quality of Life Tool (FERTIQOL). | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  The Fertility Quality of Life Tool (FERTIQOL) is used to evaluate changes in fertility related quality of life over time and to evaluate differences in fertility related quality of life between the intervention and attention control group. Self-reported fertility related quality of life is measured with this validated scale (score 0-100 with the higher, the better fertility related quality of life).
Changes in Body Mass Index (BMI) | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  Weight and height are measured according to International Standards for Anthropometric Assessment. Weight is measured when wearing light clothes and no shoes on a calibrated scale. Height is measured without shoes on a stadiometer. Weight and height allow body mass index (BMI) calculation. Changes in BMI over time and differences in BMI between the intervention and attention control group are evaluated.
Changes in waist circumference measured with a measuring tape | at baseline, 3 months, 6 months, 9 months and 12 months after randomisation
  Waist circumference is measured according to International Standards for Anthropometric Assessment with a SECA measuring tape to estimate abdominal fat. Changes in waist circumference over time and differences in waist circumference between the intervention and attention control group are evaluated.
Number of clinical pregnancies | 12 months
  Clinical pregnancy defined as evidence of a gestational sac confirmed by ultrasound. Dichotomous outcome (yes-no). Differences in number of clinical pregnancies between the intervention and attention control group are evaluated.
Time to pregnancy | 12 months
  Differences in time to pregnancy between the intervention and attention control group are evaluated.

OTHER OUTCOMES:
Use of the PreLiFe-programme assessed with app based tracking | at 3 months, 6 months, 9 months and 12 months after randomisation
  The use of the PreLiFe-programme is assessed in the intervention group by evaluating the % of participants using the PreLiFe-programme by app-based tracking.
Acceptability of the PreLiFe-programme assessed with a subscale of the Mobile App Rating Scale (MARS) | 12 months
  The acceptability of the PreLiFe-programme is assessed at the end of the study in the intervention group with a shortened version of the subjective quality subscale of the Mobile App Rating Scale (MARS)(score 0-10 with the higher the better subjective quality of the PreLiFe-programme).
Partners' support assessed with a questionnaire | at 3 months, 6 months, 9 months and 12 months after randomisation
  The partner's support during the PreLiFe-programme is assessed in the intervention group with a self-developed questionnaire to evaluate if they feel supported by their partner in maintaining a healthy lifestyle.This self-developed questionnaire is based on "The Social Support for Diet and Exercise scale of Sallis et al. (1987). It consists of 3 subscales: partners' support for diet (0-10), physical activity (0-15) and personal wellbeing (0-10), with the higher the better the partner's support.
Occurrence of adverse events | 12 months
  Differences in the occurrence of adverse events (data obtained from medical records) between the intervention and attention control group are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lie Fong, MD, PhD, Principal Investigator — KU Leuven, UZ Leuven
Locations (5):
- Belgium (5):
  - University Hospital Antwerp, Antwerp
  - Imelda Hospital Bonheiden, Bonheiden
  - Academic Hospital Sint Jan Bruges-Ostend, Bruges
  - Academic Hospital Diest, Diest
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Yes
For all the data generated during the course of this project, we will follow the prevailing standards and guidelines in documenting and depositing data sets.
  The PreLiFe research team will disseminate results from this research through presentations at public lectures, scientific institutions and meetings, and/or publication in major journals. Regarding data sharing, ICMJE recommendations will be followed.
  Individual deidentified participant data will be shared. In particular, individual participant data that underlie the results reported in our articles, after deindentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will become available from 9-36 months after the publication of the RCT-results by the PreLiFe research team.
Access Criteria: Data will only be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be shared to achieve aims in the approved proposal and for individual participant meta-analysis. Proposals should be directed to christophe.matthys@uzleuven.be (https://orcid.org/0000-0003-1770-6862). To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Boedt T, Dancet E, De Neubourg D, Vereeck S, Jan S, Van der Gucht K, Van Calster B, Spiessens C, Lie Fong S, Matthys C. A blended preconception lifestyle programme for couples undergoing IVF: lessons learned from a multicentre randomized controlled trial. Hum Reprod Open. 2023 Sep 29;2023(4):hoad036. doi: 10.1093/hropen/hoad036. eCollection 2023. PMID 38455033
- [Derived] Boedt T, Matthys C, Lie Fong S, De Neubourg D, Vereeck S, Seghers J, Van der Gucht K, Weyn B, Geerts D, Spiessens C, Dancet EAF. Systematic development of a mobile preconception lifestyle programme for couples undergoing IVF: the PreLiFe-programme. Hum Reprod. 2021 Aug 18;36(9):2493-2505. doi: 10.1093/humrep/deab166. PMID 34379119
- [Derived] Boedt T, Dancet E, Lie Fong S, Peeraer K, De Neubourg D, Pelckmans S, van de Vijver A, Seghers J, Van der Gucht K, Van Calster B, Spiessens C, Matthys C. Effectiveness of a mobile preconception lifestyle programme in couples undergoing in vitro fertilisation (IVF): the protocol for the PreLiFe randomised controlled trial (PreLiFe-RCT). BMJ Open. 2019 Jul 30;9(7):e029665. doi: 10.1136/bmjopen-2019-029665. PMID 31366659

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03790449/Prot_SAP_000.pdf